CLINICAL TRIAL: NCT05647681
Title: Analgesic Effect of a New Analgesic Based Gel(Douloff) Versus Oral Paracetamol in Acute Soft Injuries
Acronym: DOULOFF
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Monastir (Other)
Responsible Party: Principal Investigator, Pr. Semir Nouira, clinical professor, University of Monastir
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Urgence Monastir
Record Dates: First submitted 2022-12-03; First posted 2022-12-12 (Actual); Last update posted 2023-05-16 (Actual); Status verified 2023-05

CONDITIONS: Analgesia
Keywords: analgesia,topic analgesic,herbal medicine
MeSH Terms: conditions — Agnosia | interventions — Acetaminophen

STUDY DESIGN:
Intervention Model Description: multi-centre, randomized controlled trial
Who Masked: Participant, Care Provider
Masking Description: Patients are randomly assigned to receive a topic analgesic "Douloff" or palcebo associated with an oral treatment "Paracetamol" or placebo
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- topic analgesic "Douloff" (Active Comparator): Patients receive a tpic analgesic "douloff" in association with an oral treatment "placebo"
  Interventions: Drug: Douloff
- oral paracetamol (Active Comparator): Patients receive oral paracetamol in association with a topic placebo
  Interventions: Drug: paracetamol

INTERVENTIONS:
Drug: Douloff — topic gel
  Arms: topic analgesic "Douloff"
Drug: paracetamol — tablets
  Arms: oral paracetamol

SUMMARY:
Herbal medicine is commonly used to treat pain, but little is known about its effectiveness and its place in the common arsenal of analgesics .The question of whether such herbal combinations could have similar efficacy to oral analgesics in the treatment of post-traumatic soft tissue pain has not yet been investigated. Thus, we conducted this multi-center randomized controlled trial to determine the efficacy and tolerability of a new topical herbal preparation (Douloff®) compared to oral paracetamol in the treatment of acute pain secondary to soft tissue injury.

DETAILED DESCRIPTION:
Patients are eligible for enrollment if they are over 60 years of age, present to the emergency department with minor non-penetrating musculoskeletal soft tissue trauma occurring within 24 hours prior to admission to the emergency department, and require a prescription for home analgesic treatment at discharge: pain on movement (POM) with an intensity> 50 on a visual numeric scale (VNS) ranging from 0 to 10 (0 = no pain, 10 = maximum pain) Exclusion criteria are: skin lesions (dryness or excessive redness of the skin, atopic dermatitis and eczema) in the painful area, presence of a wound, joint dislocation or multiple injuries, fracture , patients with severe trauma (Injury Severity Score > 16), the need for hospitalization or surgery, daily use of NSAIDs or other analgesics in the 2 weeks before presentation, and previous treatment with analgesia for the same injury, Pregnant or lactating women , inability to use the VNS pain score, refusal to consent, or refusal to communicate Patients are ineligible if they have contraindications to any of the drugs in the protocol, including a history of previous adverse events or a known allergy or hypersensitivity.

Patients are randomly assigned (1:1) to receive Douloff or oral paracetamol.Randomization is performed centrally according to a computer-generated random list by a blinded research associate not involved in any other part of the trial. The subjects included are divided into two groups: the new gel (Douloff® group) or oral paracetamol (paracetamol group). All treatments in the protocol are numbered according to the randomization sequence by an independent research associate who is not involved in the monitoring or follow-up of the subjects. The topical study treatment is applied to the injured site 3 times daily for 7 days. The gel should be applied gently to the skin of the injured site for 1 minute. To minimize additional sources of response variability, adhesive and/or immobilizing casts, bandages, splints, and ice application are prohibited after randomization. Patients should be instructed to prevent water or moisture from contacting the affected area after application of topical therapy. Paracetamol is administered orally (1g three times daily).

The primary endpoint is the frequency of pain resolution defined as at least a 50% reduction in pain level (VNS) at day 7 compared with the ED discharge VNS (VNS D0) during movement (DAM).

Secondary end points included delta VNS, which is the change in VNS score from ED discharge (VNS D0) to 7 days later (VNS D7). The delta VNS is calculated as [(VNS D0 - VNS D7 / VNS D0) x 100]. Time to achieve pain resolution criteria, need for rescue analgesia, patient satisfaction, and rate of adverse events are also considered secondary endpoints. Failure to apply the gel more than three times during a treatment period constituted poor adherence.

ELIGIBILITY:
Inclusion Criteria:

* Patients are eligible for enrollment if they are over 60 years of age, present to the emergency department with minor non-penetrating musculoskeletal soft tissue trauma occurring within 24 hours prior to admission to the emergency department, and require a prescription for home analgesic treatment at discharge: pain on movement (POM) with an intensity> 50 on a visual numeric scale (VNS) ranging from 0 to 10 (0 = no pain, 10 = maximum pain)

Exclusion Criteria:

* Patients were excluded from the study:

If they had skin lesions (dryness or excessive redness of the skin, atopic dermatitis and eczema) in the painful area The presence of a wound, joint dislocation or multiple injuries. The presence of a fracture Patients with severe trauma (Injury Severity Score > 16) The need for hospitalization or surgery Daily use of NSAIDs or other analgesics in the 2 weeks before presentation, and previous treatment with analgesia for the same injury Contraindications to any of the drugs in the protocol, including a history of previous adverse events or a known allergy or hypersensitivity.

Pregnant or lactating women Inability to use the VNS pain score refusal to consent or communicate

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1100 (Estimated)
Dates: Start 2023-07-01 (Estimated); Primary Completion 2024-07-31 (Estimated); Study Completion 2024-07-31 (Estimated)

PRIMARY OUTCOMES:
the frequency of pain resolution defined as at least a 50% reduction in pain level (VNS) at Day 7 compared with the ED discharge VNS (VNS Day 0) during movement (DAM) | at seven days ED discharge
  resolution of pain with decrease of visual numeric scale (that range from 0: no pain to 10 :severe pain) more than 50% comparing to initial value

SECONDARY OUTCOMES:
delta VNS, which is the change in VNS score from ED discharge (VNS D0) to 7 days later (VNS D7). | at seven days ED discharge
  The delta VNS is calculated as [(VNS D0 - VNS D7 / VNS D0) x 100]
Time to achieve pain resolution | at seven days ED discharge
  time between the start of the analgesic treatment and the one when VNS (that range from 0: no pain to 10 :severe pain) decreased to less than 3.
need for rescue analgesia | at seven days ED discharge
  need for rescue analgesia
patient satisfaction | at seven days ED discharge
  Satisfaction of patients evaluated with the likert score at the ED discharge.
adverse events rate | at seven days ED discharge
  occurence of adverse events

REFERENCES:
- [Derived] Toumia M, Dhaoui R, Sassi S, Kouraichi C, Bel Haj Ali K, Sekma A, Bakir A, Jaballah R, Yaakoubi H, Youssef R, Zorgati A, Beltaief K, Mezgar Z, Khrouf M, Sghaier A, Jerbi N, Zemni I, Bouida W, Grissa MH, Saad J, Boubaker H, Boukef R, Msolli MA, Nouira S. Efficacy of a natural herbal topical analgesic versus oral paracetamol in patients with soft tissue injury: a randomized, double-blind, placebo-controlled study. Pain Med. 2025 Jun 1;26(6):329-336. doi: 10.1093/pm/pnaf006. PMID 40045174